CLINICAL TRIAL: NCT03932747
Title: Placebo-Contolled, Randomized of Creams With or Without Urea Influenceon the Hydration of the Skin of the Foot
Brief Title: Creams With or Without Urea Influence the Hydration of the Skin of the Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, PAULA COBOS MORENO, Principal Investigator, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EXAMPLE-1
Record Dates: First submitted 2019-04-08; First posted 2019-05-01 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: FOOT
Keywords: Hydration; UREA

STUDY DESIGN:
Intervention Model Description: CLINICAL TRIAL WITH THREE GROUPS: CONTROL GROUP, UREA GROUP 5% AND UREA GROUP 20%.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Creams (Placebo Comparator): Measuring the skin before the application of the cream without urea (placebo), wait 3 hours and re-measure the hydration
  Interventions: Other: pre- Hydratión skin; Other: post- Hydratión skin
- Urea 5% (Active Comparator): Measuring the skin before the application of the cream with urea (5%), wait 3 hours and re-measure the hydration
  Interventions: Other: pre- Hydratión skin; Other: post- Hydratión skin
- Urea 20% (Active Comparator): Measuring the skin before the application of the cream with urea (20%), wait 3 hours and re-measure the hydration
  Interventions: Other: pre- Hydratión skin; Other: post- Hydratión skin

INTERVENTIONS:
Other: pre- Hydratión skin — Measurement of hydration of the skin.
Other: post- Hydratión skin — Measurement of hydration of the skin.

SUMMARY:
The skin is the most external organ of our body and one of its main functions is to provide protection in terms of possible infections.

Hydration is related to the proper functioning of the skin, being more difficult the appearance of wounds or cracks, which lead to the appearance of infections or other dermatological alterations.

The skin of the feet is thicker than in the rest of the body, due to the load it supports, being more complicated to maintain it.

With this study what is intended is to assess the effectiveness of different concentrations of urea (5% and 20%) in the hydration of the foot

DETAILED DESCRIPTION:
The measuring device of the Corneometer is constituted by a cylindrical probe, which contains at its distal end two parallel circuits in the form of capacitors covered by a plastic membrane. The probe should be placed perpendicularly on the surface of the skin. The pressure exerted on it must always be the same, therefore the probe has an internal hydraulic mechanism that, regardless of the pressure exerted by the manipulator, maintains a constant pressure.

Once the probe is placed in the place of measurement and the pressure is exerted on the skin, the circuit is closed and the conductance or capacitance is determined depending on the device, in a fraction of a second. Usually, between 3 and 10 measurements are made for each determination and entered in a computer record to obtain their averages.

The capacity of the condenser depends on the material, most of the materials increase the capacity compared to the vacuum by a factor of more than seven (dielectric constant); Water, however, increases the capacity by a factor of 81. Therefore, variations in the water content in the skin produce strong modifications in the measuring range of the Corneometer CM 825.

The Corneometer uses relative units proportional to the degree of corneal wetting. One AU corresponds to 0.2-0.9 mg of water per mg of anhydrous stratum corneum.

The study will be carried out to young people (20 -26 years old) from Practicum I of the Podiatry Clinic University of Plasencia.

The inclusion criteria will be those people who want to voluntarily participate in the study.

Those who suffer from structural, functional or traumatic alterations that affect the morphology and function of the lower limb, disorders that affect the skin, wounds, blisters are excluded from the study. Those who do not fall within the age range of the study and who have used creams or any type of lotion the night before on the feet are also excluded.

First, three randomized groups are performed, since each group will be treated with a different cream: placebo, 5% urea cream and 20% cream. The investigator will be blinded as well as the patients, since neither will know what cream is being applied.

Secondly, the subjects participating in the study will be explained, the objectives of the study and that for this need to perform a test using a non-invasive instrument that allows us to detect the superficial hydration of participants skin.

Thirdly, instructed to sign the informed consent, if so, participants are asked to accompany us to a previously heated room and be accommodated in the podiatric chair.

Subsequently, the patient is asked to answer some questions (Age, Name and surname). In addition, the researcher will note the temperature and humidity in which the room is located and the presence of hyperkeratosis on the sole of the patient's foot and area of appearance. (Annex 3)

Finally, before proceeding to the measurement, the patient is positioned barefoot with the legs stretched over the legs, then the researcher passes a gauze impregnated in alcohol of 70% to eliminate possible remains that could interfere with the measurement.

After checking that the alcohol has evaporated, explore the sole of the foot and mark on our data collection sheet, if at the points where participants are going to measure there is a presence or not of hyperkeratosis.

In this case is going to measure 3 points of each foot that are:

* First metatarsal head
* Fifth metatarsal head
* Heel

These points are considered important because they serve as support for the foot when the subject is standing, since they form the three basic points of foot support.

To carry out the hydration measurement, the investigators place the probe or head of the Corneometer on the surface of the skin and exert pressure until the appearance of an acoustic signal that indicates that the measurement has been recorded. This process is done 3 times in each zone that they want to measure to obtain 3 records and thus reduce the margin of error derived from the measurement.

To finish, the investigators will apply cream (placebo, urea 5% or 20%) depending on the study group to which it belongs, and they will fit him and the investigators will measure again in about three hours, taking the hydration of the three points mentioned above.

Once all the data of the participants have been registered, and the measurements coming from the hydration, the resulting values are analyzed.

ELIGIBILITY:
Inclusion Criteria:

* those people who want to voluntarily participate in the study.

Exclusion Criteria:

* suffer from structural, functional or traumatic alterations that affect the morphology and function of the lower limb
* who do not fall within the age range of the study
* who have used creams or any type of lotion the night before on the feet

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Pre-hydration of the study areas | 5 minutes
  Measurement of the hydration of the three study areas (first metatarsal head, fifth metatarsal head and heel). The measure that the corneometer gives us is UA (water per mg stratum corneum)
Pre and Post of all study areas | 5 MINUTES
  Measurement of the hydration of the three study areas (first metatarsal head, fifth metatarsal head and heel) after the application of the different creams. The measure that the corneometer gives us is UA (water per mg stratum corneum).
Comparison of hydration of study areas in placebo vs. 5% groups as determined using corneometer UA (water per mg stratum corneum) | 3 hours after the application
  It is compared if the hydration of the different study areas depending on the type of cream that has been used.
Comparison of hydration of study areas in placebo vs. 20% groups as determined using corneometer UA (water per mg stratum corneum) | 3 hours after the application
  It is compared if the hydration of the different study areas depending on the type of cream that has been used.
Comparison of hydration of study areas in 20% vs. 5% groups as determined using corneometer UA (water per mg stratum corneum) | 3 hours after the application
  It is compared if the hydration of the different study areas depending on the type of cream that has been used.

CONTACTS AND LOCATIONS:
Overall Officials: BEATRIZ GOMEZ MARTIN, PODOLOGÍA, Study Director — CENTRO UNIVERSITARIO DE PLASENCIA
Locations (1):
- Centro Universitario de Plasencia, Plasencia, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No